CLINICAL TRIAL: NCT06734780
Title: Effects of Vaping on Post-operative Recurrence of Crohn's Disease: a Retrospective Multicenter Study
Brief Title: Effects of Vaping on Post-operative Recurrence of Crohn's Disease
Acronym: VAPE-CD
Status: Recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Tommaso Lorenzo Parigi, MD Gastroenterologist, IRCCS Ospedale San Raffaele
Other Study IDs: VAPE-CD
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-08

CONDITIONS: The Impact of Vaping on Crohn's Disease Endoscopic Recurrence After Resection
Keywords: Crohn; e-cigarette; smoke; tobacco; heat-not-burn tobacco; postoperative recurrence
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients (age ≥18) diagnosed with CD: Patients who underwent intestinal resections due to Crohn's disease or its complications

SUMMARY:
Tobacco smoke is a well-established risk factor for post-operative recurrence of Crohn's disease. Over the last few decades electronic cigarettes have gained popularity as an alternative to traditional tobacco, however, their effects on Crohn's disease are unknown.

Tobacco smoke negatively impacts most outcomes of Crohn's disease including, but not limited to, response to therapy and risk of hospitalization. Smoke is particularly relevant in the post-operative setting, as it increases the chance of disease recurrence after surgical resection, and therefore prophylactic treatment with biologics is recommended in Crohn's patients who smoke.

At present, there are no studies evaluating the impact of e-cigarette smoke on post-operative recurrence and therefore informing physicians on the appropriateness of prophylactic treatment in this subset of patients. This study aims to assess the impact of vaping (or smoking of electronic cigarettes) on Crohn's disease endoscopic recurrence after resection as compared to non-smoke and smoke of traditional tobacco cigarettes.

DETAILED DESCRIPTION:
This is a multicenter study with the aim of evaluate the effect of e-cigarette smoke (vaping) on Crohn's disease post-operative. Secondary objectives are :

* To evaluate the effect of e-cigarette smoke on Crohn's disease postoperative recurrence compared to tobacco smoke.
* To determine the effect of heat-not-burn tobacco products (ie. IQOS) on Crohn's disease postoperative recurrence compared to tobacco smoke.
* To determine the effect of tobacco smoke on Crohn's disease postoperative recurrence compared to nonsmokers.
* To account for the confounding effect of known risk factors of post- operative recurrence: biologic treatment for postoperative prophylaxis, penetrating complications, multiple intestinal resections.

The subjects considered are adult patients (≥18 years) diagnosed with CD who underwent surgical resections of a tract of intestine accessible through endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥18) patients with an established diagnosis of Crohn's disease.- Patients who underwent surgical resections of a tract of intestine accessible through endoscopy.
* Patients who underwent ileo-colic resections due to Crohn's disease or its complications (stricture or fistula) irrespective of the type of anastomosis (side-to-side L-L, , end-to-end T-T, end-to-side T-L, Kono S, iso or antiperistaltic)
* Patients whose smoking habit (or nonsmoking habit) is clearly reported in the medical records
* Data will be collected from January 2000 to August 2024.

Exclusion Criteria:

* Patients who underwent surgical operations different from intestinal resections (i.e. stricturoplasty raffias, dilation, bypass etc)
* Patients who underwent Intestinal resections for indications other than Crohn's disease (inflammatory, stricturing or fistulizing) such as: cancer, trauma, etc
* Patients who for any reason did not undergo endoscopic reassessment of the anastomosis within 12 months from surgery
* Unconfirmed diagnosis of Crohn's disease
* Patients whose smoking habits could not be determined
* Patients with mixed smoking habits, defined as smoking at the same time tobacco cigarettes and e-cigarettes or who have changed type of smoking product (from tobacco to vaping or vice versa) after the intestinal resection and before the endoscopic reassessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (age ≥18) patients with an established diagnosis of Crohn's disease who underwent surgical resections of a tract of intestine accessible through endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Endoscopic recurrence e-cigarettes vs no-smoke | Endoscopic recurrence will assessed within the first 12 months after an intestinal surgical resection for active or complicated Crohn's disease.
  Rate of endoscopic recurrence (defined as a Rutgeerts score ≥ i2) in patients who smoke e-cigarettes in the first year after intestinal resection for active Crohn's disease compared to the endoscopic recurrence rate in patients who do not smoke.

SECONDARY OUTCOMES:
Endoscopic recurrence e-cigarettes vs tobacco | Endoscopic recurrence assessed within the first 12 months after an intestinal surgical resection for active or complicated Crohn's disease.
  The rate of endoscopic recurrence (defined as a Rutgeerts score ≥i2) in patients who smoke e-cigarettes in the first year after an intestinal resection for active Crohn's disease compared to the endoscopic recurrence rate in patients who smoke tobacco cigarettes.
Endoscopic recurrence tobacco vs no-smoke | Endoscopic recurrence assessed within the first 12 months after an intestinal surgical resection for active or complicated Crohn's disease.
  The rate of endoscopic recurrence (defined as a Rutgeerts score ≥i2) in patients who smoke tobacco cigarettes in the first year after an intestinal resection for active Crohn's disease compared to the endoscopic recurrence rate in patients who do not smoke.
Endoscopic recurrence heat-not-burn tobacco vs tobacco | Endoscopic recurrence assessed within the first 12 months after an intestinal surgical resection for active or complicated Crohn's disease.
  The rate of endoscopic recurrence (defined as a Rutgeerts score ≥i2) in patients who smoke heat-not-burn tobacco products in the first year after an intestinal resection for active Crohn's disease compared to the endoscopic recurrence rate in patients who smoke tobacco cigarettes.
Risk of recurrence | Endoscopic recurrence assessed within the first 12 months after an intestinal surgical resection for active or complicated Crohn's disease.
  Odds ratio of endoscopic recurrence between e-cigarettes and non-smokers calculated with a multivariable logistic regression analysis including the following variables: biologic prophylactic treatment, intestinal resections prior to index surgery, penetrating complications

CONTACTS AND LOCATIONS:
Overall Officials: Tommaso Lo Parigi, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Michigan, Italy

IPD SHARING:
Plan to Share IPD: No